CLINICAL TRIAL: NCT06027307
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Effects of Enavogliflozin on Outcomes in Patients With Functional Tricuspid Regurgitation and Heart Failure With Preserved Left Ventricular Ejection Fraction
Brief Title: Enavogliflozin Outcome Trial in Functional Tricuspid Regurgitation
Acronym: EVENT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-0070
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Tricuspid Regurgitation; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Tricuspid Valve Insufficiency | interventions — Enavogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enavogliflozin (Experimental): Enavogliflozin 0.3 mg qd for 18 months
  Interventions: Drug: Enavogliflozin
- Placebo (Placebo Comparator): Placebo qd for 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enavogliflozin — All study patients will receive enavogliflozin in addition to their prior medications. They will receive optimal medical treatment for their underlying disease such as hypertension, diabetes, arrhythmia and/or coronary artery disease.
  Other Names: Envlo (brand name)
  Arms: Enavogliflozin
Drug: Placebo — All study patients will receive placebo in addition to their prior medications. They will receive optimal medical treatment for their underlying disease such as hypertension, diabetes, arrhythmia and/or coronary artery disease.
  Arms: Placebo

SUMMARY:
The Enavogliflozin Outcome Trial in Functional Tricuspid Regurgitation (EVENT) was designed to examine the hypothesis that, compared with placebo, therapy with the SGLT2 inhibitor enavogliflozin would improve clinical and echocardiographic outcomes in heart failure (HF) patients with functional tricuspid regurgitation (TR) and preserved left ventricular ejection fraction (LVEF).

The primary objective of the EVENT study is to test the hypothesis that, compared with placebo, therapy with enavogliflozin for 18 months would improve a composite of cardiovascular events or worsening of TR on follow-up echocardiography in HF patients with functional TR and preserved LVEF. The secondary objective is to examine whether enavogliflozin is effective in reduction of renal events and tricuspid regurgitation, and to evaluate whether beneficial effects of enavogliflozin on primary outcomes are associated with reduction of all-cause mortality.

DETAILED DESCRIPTION:
Functional tricuspid regurgitation (TR) develops due to functional and structural alterations related to heart failure (HF), mitral valve disease and atrial fibrillation. An increase in cardiac filling pressure due to left ventricular (LV) systolic or diastolic dysfunction leads to left atrial, right atrial (RA) and right ventricular (RV) remodeling, which causes tricuspid annular dilatation and TR. The development of significant functional TR causes RV dysfunction and further dilation of RV, which deteriorates TR. Functional TR may occur with HF with preserved or reduced ejection fraction (EF), and the prevalence of moderate-to-severe functional TR is around 19% in patients with HF. Regardless of LVEF or pulmonary artery pressure, presence of moderate or severe functional TR is associated with more symptoms, reduced cardiac output, and worse renal function. A vicious cycle of significant TR, RV volume overload, adverse remodeling of RA, RV, and tricuspid annulus, and consequent aggravation of TR is suggested as a pathophysiologic mechanism of the poor clinical outcomes of patients with TR, and the presence of moderate or severe functional TR is a strong independent determinant of mortality in patients with HF. Because functional TR has a strong prognostic impact and plays an important pathophysiologic role in patients with HF, functional TR is suggested as a therapeutic target in HF. However, there have been no proven medical therapies for TR and only loop diuretics are cautiously recommended for relief of congestive symptoms in patients with severe TR and signs of RV failure. In patients with functional TR associated with systolic dysfunction, medical therapy for HF with a reduced EF may diminish functional TR by improving LV systolic function. Otherwise, the morbidity and mortality of patients with functional TR remain high and a novel therapeutic agent is needed to improve clinical outcomes of HF patients with functional TR and a preserved LV ejection fraction.

Sodium-glucose co-transporter 2 (SGLT2) inhibitors induce urinary excretion of glucose and sodium by blocking the SGLT2 transporter in the proximal tubule (8). SGLT2 inhibitor-induced natriuresis lower cardiac preload and reduce pulmonary congestion and systemic edema. SGLT2 inhibitors also restore tubuloglomerular feedback and lower the intraglomerular pressure by vasoconstriction of the afferent arterioles and consequently reduce hyperfiltration-related renal damage. The beneficial effects of SGLT2 inhibitors on the heart and kidneys may halt the vicious cardiorenal cycle in patients with functional TR (9), which results in deterioration of renal function, hospitalization for heart failure, and cardiovascular mortality.

Accordingly, the Enavogliflozin Outcome Trial in Functional Tricuspid Regurgitation (EVENT) will test the hypothesis that, compared with placebo, therapy with the SGLT2 inhibitor enavogliflozin for 18 months would improve clinical and echocardiographic outcomes in HF patients with functional TR and preserved LVEF.

ELIGIBILITY:
Inclusion Criteria:

* Patients must agree to the study protocol and provide written informed consent
* Outpatients male or female between the age of 20 and 80
* Non-diabetic or type2 DM patients with HbA1c 6.5-10.5%
* HF with dyspnea of NYHA functional class II or III
* Presence of moderate or severe functional TR and preserved LVEF on echocardiography

  * TR whose vena contracta ≥ 0.3cm, effective regurgitant orifice area ≥ 0.20 cm2, or jet area > 10cm2
  * LVEF ≥ 50%
* NT-proBNP >125 pg/mL or BNP ≥35 pg/mL

Exclusion Criteria:

* History of hypersensitivity or allergy to the study drugs, drugs of similar chemical classes, as well as known or suspected contraindications to the study drug
* Current use or prior use of a SGLT-2 inhibitor or combined SGLT-1 and 2 inhibitor
* Any evidence of structural tricuspid valve disease
* Any significant left-sided valve disease
* Left ventricular ejection fraction <50%
* Marked bradycardia or 2nd or 3rd degree AV block
* Intracardiac devices (CRT, ICD, Pacemaker)
* Hypertrophic or restrictive cardiomyopathy
* Severe pulmonary hypertension: TR Vmax > 3.5m/s at screening
* Medical history of hospitalization within 4 weeks
* Current acute decompensated heart failure or dyspnea of NYHA functional class IV
* Symptomatic hypotension and/or a SBP < 90 mmHg at screening
* Uncontrolled hypertension (SBP≥180mmHg or DBP≥110mmHg)
* Estimated GFR < 30 mL/min/1.73m2
* History of ketoacidosis
* Evidence of hepatic disease as determined by any one of the following: AST or ALT values exceeding 2 x upper limit of normal (ULN) at screening visit (Visit 0), history of hepatic encephalopathy, history of esophageal varices, or history of portocaval shunt.
* Acute coronary syndrome, stroke, major CV surgery, PCI within 3 months
* Plan for cardiac surgery, PCI or ablation of atrial flutter of fibrillation
* History of severe pulmonary disease
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using a barrier method plus a hormonal method
* Pregnant or nursing (lactating) women
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the investigator, would preclude safe completion of the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular event | 18 months
  A composite of cardiovascular death, hospitalization for HF, or worsening of tricuspid regurgitation that occurs during follow-up

SECONDARY OUTCOMES:
All-cause death | 18 months
  All-cause death occurring during follow-up
Cardiovascular clinical event | 18 months
  A cardiovascular composite (cardiovascular mortality or hospitalization for HF) occurring during follow-up
Renal event | 18 months
  A renal composite (doubling of serum creatinine, decrease in the eGFR of 30% or more, renal replacement therapy, or renal death) occurring during follow-up
Change of TR | 18 months
  Change of TR on echocardiography from baseline to 18 months follow-up
Change of RV strain | 18 months
  Change of RV strain on echocardiography from baseline to 18 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: DUK HYUN KANG, MD, Principal Investigator — Asan Medical Center
Locations (5):
- South Korea (5):
  - Inha University Hospital, Incheon
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No